CLINICAL TRIAL: NCT00861146
Title: Concurrent Alcohol and Smoking Treatment: Effects on Alcohol Relapse Risk
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0804003723; R01AA011197 (NIH)
Record Dates: First submitted 2009-03-11; First posted 2009-03-13 (Estimated); Results first posted 2014-04-07 (Estimated); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Tobacco Use Cessation; Alcohol-related Disorders
Keywords: nicotine dependence; tobacco dependence; smoking cessation; alcoholism; self-efficacy; relapse
MeSH Terms: conditions — Tobacco Use Cessation; Alcohol-Related Disorders; Tobacco Use Disorder; Smoking Cessation; Alcoholism; Recurrence | interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 concurrent smoking cessation (Experimental): smoking cessation delivered concurrent with intensive alcohol treatment
  Interventions: Behavioral: behavioral counseling plus contingency management
- 2 deferred smoking cessation (Active Comparator): smoking cessation delivered 12 weeks after intensive alcohol treatment
  Interventions: Behavioral: behavioral counseling plus contingency management

INTERVENTIONS:
Behavioral: behavioral counseling plus contingency management — Individual counseling sessions with voucher rewards for smoking abstinence, transdermal nicotine patch and nicotine gum

SUMMARY:
The majority of individuals with alcohol problems remain current smokers, and the negative health consequences of smoking among these individuals are substantial. This study will investigate the impact of smoking cessation interventions initiated during intensive alcohol treatment on processes reflecting risk of alcohol relapse.

DETAILED DESCRIPTION:
Objectives:

Most alcohol and drug treatment programs do not systematically address cigarette smoking during treatment. One obstacle is a concern that smoking cessation early in recovery might increase risk of alcohol relapse. This study followed patients enrolled in intensive outpatient alcohol treatment to compare the effects of a Concurrent Smoking Cessation (CSC) intervention to a Deferred Smoking Cessation (DSC) control group on process measures reflecting risk of alcohol relapse.

Research Design:

Participants were enrolled in intensive outpatient alcohol treatment and then randomized to CSC or DSC groups in a 2:1 ratio. The CSC group received smoking treatment concurrent with intensive alcohol treatment and the DSC group received smoking treatment three months after alcohol treatment. The smoking treatment protocol included behavioral counseling, contingency management with voucher rewards for verified smoking abstinence, and prescribed nicotine patch and gum. During a three-month period after the CSC target smoking quit date, both groups of subjects were asked to participate in a prospective daily monitoring procedure, calling into an Interactive Voice Response system once a day to complete self-report assessments of relapse risk factors. By comparing participants in the CSC group composed of many participants who have stopped smoking with the DSC group who are expected to continue smoking during this daily monitoring period, we will determine the impact of smoking cessation on alcohol relapse risk factors.

Methodology:

This study was conducted in the substance abuse day treatment programs located at Newington and West Haven campuses of VA Connecticut Healthcare System. These are three-week treatment programs meeting Monday-Friday for 4-5 hrs/day. Participants were recruited either before or soon after day program admission. Participants 151 individuals that are 18 years of age or older, meet Diagnostic and Statistical Manual-IV (DSM-IV) criteria for current alcohol abuse or dependence, report currently smoking 1 or more cigarettes per day, and are screened for medical contraindications for nicotine patch and gum use. Dependent variables are process assessments reflecting alcohol relapse risk obtained using daily Interactive Voice Response (IVR) technology. These relapse risk processes include alcohol craving, negative affect, alcohol abstinence self efficacy, alcohol outcome expectancies, motivation for alcohol abstinence, and self-control demands. Given the mixed results from previous clinical trials, we conducted bidirectional tests of the hypothesis that smoking cessation has an impact on alcohol relapse risk factors, examining whether smoking cessation leads to increased or decreased alcohol relapse risk.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV criteria for alcohol abuse or dependence
* Age 18 or older
* English speaking
* Smoking 1 or more cigarettes/day
* Male or female veterans eligible for VA healthcare
* Female nonveterans also eligible

Exclusion Criteria:

* Allergy or hypersensitivity to nicotine or adhesives used in nicotine patch
* Weigh less than 100 lbs
* Lack of interest in stopping smoking
* Pregnant or lactating females or females not practicing acceptable form of contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2009-04; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ned L Cooney, PhD, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - VA Connecticut Healthcare System, Newington, Connecticut
  - VA Connecticut Healthcare System, West Haven, Connecticut

REFERENCES:
- [Derived] Cooney NL, Litt MD, Sevarino KA, Levy L, Kranitz LS, Sackler H, Cooney JL. Concurrent alcohol and tobacco treatment: Effect on daily process measures of alcohol relapse risk. J Consult Clin Psychol. 2015 Apr;83(2):346-58. doi: 10.1037/a0038633. Epub 2015 Jan 26. PMID 25622198

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment May 2009 to October 2012.
  Excluded (n=1448):
  Does not smoke, does not drink (n=678) Declined to participate (n=320) Medical problems (n=297) Otherwise ineligible (n=112) Male non-vet (n=41)
Period: Overall Study
Arm/Group | 1 Concurrent Smoking Cessation | 2 Deferred Smoking Cessation
Started | 105 | 46
Week 2 Assessment | 97 | 45
Week 13 Assessment | 85 | 38
Completed | 85 | 38
Not Completed | 20 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 Concurrent Smoking Cessation | 2 Deferred Smoking Cessation | Total
Number analyzed (Participants) | 105 | 46 | 151
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.5 (9.07) | 48.1 (8.68) | 49.1 (8.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 7 | 21
  Male | 91 | 39 | 130
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 43 | 20 | 63
  White | 57 | 25 | 82
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 1 | 6
Region of Enrollment [Number; unit: participants]
  United States | 105 | 46 | 151
Cigarettes smoked/day [Mean (Standard Deviation); unit: cigarettes] | 16.0 (8.0) | 16.8 (10.0) | 16.2 (8.7)
Proportion days heavy drinking [Mean (Standard Deviation); unit: proportion] — Heavy drinking days were defined as days with > 6 standard drinks per day for men and > 4 standard drinks per day for women. The baseline measure examined the proportion of heavy drinking days in the 90 days prior to the last day of reported drinking prior to study enrollment.
  proportion | .58 (.33) | .52 (.38) | .56 (.35)

OUTCOME MEASURES:

1. Primary Outcome: Smoking Abstinence
Description: 7-day point prevalence smoking abstinence verified by breath carbon monoxide missing coded as smoking
Time Frame: 12 weeks
Measure: Number; unit: participants
Arm/Group | 1 Concurrent Smoking Cessation | 2 Deferred Smoking Cessation
Number analyzed (Participants) | 105 | 46
participants | 20 | 1
Statistical Analysis 1: Comparison: 1 Concurrent Smoking Cessation vs 2 Deferred Smoking Cessation; Test type: Superiority or Other; p < .01, Chi-squared; df = 1

2. Secondary Outcome: Proportion of Days Heavy Drinking
Description: Heavy drinking days were defined as days with > 6 standard drinks per day for men and > 4 standard drinks per day for women. This measure examined the proportion of days heavy drinking across 28 days in follow-up weeks 9-12.
Time Frame: follow-up weeks 9-12
Measure: Mean (Standard Deviation); unit: proportion of days
Arm/Group | 1 Concurrent Smoking Cessation | 2 Deferred Smoking Cessation
Number analyzed (Participants) | 85 | 38
proportion of days | .0332 (.1130) | .0132 (.0375)
Statistical Analysis 1: Comparison: 1 Concurrent Smoking Cessation vs 2 Deferred Smoking Cessation; Drinking outcomes assessed using the timeline follow-back were evaluated with mixed model regression analyses using maximum likelihood estimation. Time was measured in three monthly periods and treated as a repeated factor (due to the fixed time period between estimates); Test type: Superiority or Other; p > .15, mixed model regression analyses; mixed model regression analyses (F) = 2.04

3. Primary Outcome: Smoking Abstinence
Description: 7-day point prevalence smoking abstinence verified by breath carbon monoxide missing coded as smoking
Time Frame: 2 weeks
Measure: Number; unit: participants
Arm/Group | 1 Concurrent Smoking Cessation | 2 Deferred Smoking Cessation
Number analyzed (Participants) | 105 | 46
participants | 53 | 1
Statistical Analysis 1: Comparison: 1 Concurrent Smoking Cessation vs 2 Deferred Smoking Cessation; Test type: Superiority or Other; p < .001, Chi-squared; df=1

ADVERSE EVENTS:
Arm/Group | 1 Concurrent Smoking Cessation | 2 Deferred Smoking Cessation
Serious Adverse Events (participants affected / at risk) | 4/105 | 2/46
Other Adverse Events (participants affected / at risk) | 60/105 | 12/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 Concurrent Smoking Cessation (N=105) | 2 Deferred Smoking Cessation (N=46)
Hospitalization psychiatric (Psychiatric disorders) | 2 (2) | 1 (1) — unrelated
Hospitalization alcohol (Psychiatric disorders) | 1 (1) | 0 (0) — unrelated
Hospitalization stroke (Nervous system disorders) | 1 (1) | 1 (1) — unrelated
Hospitalization gastrointestinal (Gastrointestinal disorders) | 0 (0) | 1 (1) — unrelated
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 Concurrent Smoking Cessation (N=105) | 2 Deferred Smoking Cessation (N=46)
vivid dreams (Psychiatric disorders) | 32 (32) | 7 (7)
itching or irritation (Skin and subcutaneous tissue disorders) | 30 (30) | 5 (5)
dry mouth (Gastrointestinal disorders) | 19 (19) | 3 (3)
coughing (Respiratory, thoracic and mediastinal disorders) | 14 (14) | 3 (3)
insomnia (Psychiatric disorders) | 8 (8) | 1 (1)
heartburn or indigestion (Gastrointestinal disorders) | 8 (8) | 1 (1)
rash (Skin and subcutaneous tissue disorders) | 7 (7) | 2 (2)
hiccups (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No